CLINICAL TRIAL: NCT06797011
Title: Efficacy of Plasmapheresis in Patients of Drug-Induced Liver Injury (DILI) With Underlying Chronic Liver Disease: An Open Labelled RCT
Brief Title: Efficacy of Plasmapheresis in Patients of Drug-Induced Liver Injury (DILI) With Underlying Chronic Liver Disease
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-DILI-01
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Drug Induced Liver Injury; Chronic Liver Disease
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLEX with SMT (Experimental): High Volume Plex with minimum 3 sessions on alternate days along with Standard treatment.
  Interventions: Biological: High volume Plasma Exchange; Other: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Standard treatment.
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: High volume Plasma Exchange — High volume Plasma Exchange with minimum 3 sessions on alternate days
  Arms: PLEX with SMT
Other: Standard Medical Treatment — Standard Medical Treatment includes stopping the offending drug,nutrition,injection NAC,Tablet UDCA,steroid in DILI AIH

SUMMARY:
DILI is an underdiagnosed and under appreciated causal or contributing factor to liver injury. DILI can mimics features of the entire spectrum of acute and chronic liver disease.

Asia-Pacifc region is characterized by two unique features; the high prevalence of tuberculosis (TB) in the population and the ubiquitous use of traditional and complimentary medicines.Current definition of Hy's law presents significant difficulties when dealing with patients with preexisting CLD in clinical trials. Hallmark of the hepatic manifestation in these patients is hyperbilirubinemia and coagulopathy rather than ALT elevation.

DETAILED DESCRIPTION:
Study Design Single-center, non-blinded, parallel group, randomized controlled trial. Allocation ratio between two groups: 1:1.

Study population: Adults aged 18-75 years with previously known or unknown underlying CLD Diagnosis of DILI-based causality of assessment by RECAM. Severe DILI with bilirubin > 12mg/dl or INR>2, S.Bili >5 mg/dl Consent to participate in the study (based on biopsy, imaging or clinical criteria).

Study design: RCT Study period: 1 year Sample size: 96 Intervention: Patients after screening for all exclusion criteria will be randomized into either the standard treatment group or the plasma exchange group.

Monitoring and assessment: All patients would undergo vital and baseline parameter screening before randomization. Based on randomization they will receive either steroid or plasma exchange followed by steroid.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-75 years with previously known or unknown underlying CLD.
2. Diagnosis of DILI based causality of assessment by RECAM.
3. Severe DILI with bilirubin > 12mg/dl or INR>2, S.Bili >5 mg/dl.
4. Consent to participate in the study (based on biopsy/imaging/or clinical criteria).

Exclusion Criteria:

1. Active infection
2. Contraindications to plasmapheresis (e.g., severe coagulopathy, hemodynamic instability, patients with sepsis, shock, poor P/F ratio).
3. Pregnant or breastfeeding women.
4. HCC or any malignancy
5. UGI bleed, uncontrolled HE
6. Option LTx being considered
7. S. Creatinine > 2mg/dL
8. DILI ALF
9. Alcoholic Hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Liver Transplant free survival at the end of 30 days between two groups. | 30 days

SECONDARY OUTCOMES:
Changes in arterial lactate levels, on lactate clearance at 0, 3, 5 days | 0, 3, 5 days
Reduction in von Willebrand factor levels, endothelial function, and coagulopathy at 0 and 30 day. | 0 and 30 day.
Changes in the inflammatory milieu, IL6, IL10, and TNF alpha at 0 and 30 day. | 0 and 30 day.
Change in liver-related decompensation events (ascites, HE, variceal bleed) at 0, 3, 5,30, and 90 days. | 0, 3, 5,30, and 90 days.
Change in serum bilirubin and bile acids clearance at 0, 3, 5,30 and 90 days. | 0, 3, 5,30 and 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided